CLINICAL TRIAL: NCT03765853
Title: Randomized Study on the Evaluation of the Regular Practice of Standardized Postures Stretching Postural® in Secondary Prevention of Low Back Pains During Pregnancy.
Acronym: GEMALODO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-50; 2018-A01759-46 (Other: ID RCB)
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching Postural® (Other)
  Interventions: Other: Physiotherapy
- Control (No Intervention)

INTERVENTIONS:
Other: Physiotherapy — Usual prevention methods (ergonomic education) and Stretching Postural® postures.
  Arms: Stretching Postural®

SUMMARY:
Lower back pain (LBP) during pregnancy is a frequent syndrome: it concerns two thirds of pregnant women. This complaint isn't routinely searched for and therefore underdiagnosed. Furthermore, few solutions are given to these women in order to reduce their pain, and indirectly to improve everyday life. What's more, LBP is the cause of many work interruptions. Physical exercise during pregnancy is recommended by the National College of Gynaecologists and Obstetricians for low risk pregnancies. Several techniques have proven to be efficient.

The main objective of our study is to assess the benefit of regular practice of standardised Stretching Postural® postures in patients presenting "de novo" lower back pain during pregnancy.

The Stretching Postural® technique comprises of static postures involving muscular contractions and stretches. This allows the strengthening of the postural muscles, including the paravertebral muscles. After a short learning period, postures can be done autonomously by the patients. The postures are adaptable to each and everyone's morphology and physical limitations.

Our study is an open, prospective, randomised monocentric superiority trial in parallel branches involving major patients during low risk pregnancies. These women suffer from "de novo" lower back pain during the second and third trimesters of their pregnancies. Each patient will be randomly assigned to one of the following 2 groups:

* Stretching Postural® group (group A): usual prevention methods (ergonomic education) and Stretching Postural® postures.
* "Control" group (group B): usual prevention methods only.

Patients presenting "de novo" LBP are included in the study after a routine consult then randomly separated into two groups. During the initial consult, the physician assesses inclusion and judgement criteria, collects informed consent from the patients and teaches them the usual prevention methods as well as, concerning group A, Stretching Postural® postures. Computerized support agendas are given in order to improve observance.

Patients are evaluated at day 0 (initial evaluation), after 4 weeks (intermediate) and after 8 weeks (final), according to the main judgment criterion, as well as on secondary pain criteria by the Concise Pain Questionnaire, on their quality of life, the rate of work interruptions and their satisfaction rate. Neonatal outcome is collected at birth. Intermediate phone interviews will allow psychological support and improve observance. Inclusion is scheduled to last 22 months; each subject will be followed during a period of 2 months. The total duration of the study is 2 years.

Expected results are a decrease in back pain and an improvement of the quality of life in group A. Decrease in pain scale, equivalent to overall pain during the last week between the two groups will be our main judgment criterion. In order to detect a difference of 1.5 pain scale points (on a scale from 1 to 10) with an alpha risk of 5%, 80% magnitude and a standard deviation of 2, 56 subjects are necessary; 28 in each group.

Perspectives: This study will allow for a better diagnosis of lower back pain during pregnancy, and, consequently, for the implementation of routine means of care such as collective or private lessons in Stretching Postural® and the supply of personalised prevention documents.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients between 15 and 32 amenorrhea at the beginning of the study
* Absence of pre existing major lower back pain
* Back or lumbar pain and/or sacroiliac
* Good understanding of French
* BMI before pregnancy <35
* singletons
* Low risk pregnancy : no maternal and foetal major pathology (absence of professional risk, no antecedent of obstetric pathology, major gynecological pathology, exposure to toxic, important medical risk factors, infectious disease)
* Possibility to listen a computer audio
* Patient having accepted to participate to the study and having signed informed consent.

Exclusion Criteria:

* Physical handicap not allowing the change of positions in autonomy
* Severe cardiac, lung,hepatic, rheumatological pathology
* Sciatic without LPB (Low Back Pain), motor deficit or slipped disc
* High risk pregnancy
* maternal plan : antecedent of late miscarriage, cervix cerclage, disease having an impact on pregnancy, unbalanced diabetes insulin.
* foetal plan : multiple pregnancy, severe intrauterine growth retardation, severe foetal pathology.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Change in Lower Back Pain | 2 months
  Evaluated on the Numeric Pain Rating Scale (0 = No pain to 10 = Worst possible pain). This scale, validated, is a self-assessment of the average pain felt during the last week collecting by an evaluation questionnaire. It's part of Concise Pain Questionnaire's questions.

SECONDARY OUTCOMES:
Assessment of the analgesic efficacity on the Numeric Pain Rating Scale representing the average pain on the last week at 4 weeks. | week 4
  Evaluated on the Numeric Pain Rating Scale (0 = No pain to 10 = Worst possible pain). Questionnaire will be completed during intermediate consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier Arnaud, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Service de Gynécologie Obstétrique - Hôpital Nord, Marseille, Marseille Cedex, France